CLINICAL TRIAL: NCT07047300
Title: Effect of Heel Lift Insole on Kinematics and Kinetics of the Lower Limb and Lumbar Spine Among Healthy Individuals
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Abdelrahman Salah Sawan, Teaching assistant, Cairo University
Other Study IDs: P.T.REC/012/005801
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Healthy Individuals
Keywords: Heel Lift Insole; Electromyography (EMG); Kinetics; Kinematics; Lower Limb; Lumbar spine; Kinovea software

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Males Group (Group A)
  Interventions: Diagnostic Test: Record EMG maximum amplitude from bilateral erector spinae, rectus femoris, and medial and lateral gastrocnemius muscles.; Diagnostic Test: Photograph participants from anterior and lateral views to assess knee valgus angle and lumbosacral angle.
- Females Group (Group B)
  Interventions: Diagnostic Test: Record EMG maximum amplitude from bilateral erector spinae, rectus femoris, and medial and lateral gastrocnemius muscles.; Diagnostic Test: Photograph participants from anterior and lateral views to assess knee valgus angle and lumbosacral angle.

INTERVENTIONS:
Diagnostic Test: Record EMG maximum amplitude from bilateral erector spinae, rectus femoris, and medial and lateral gastrocnemius muscles. — Conduct measurements under two conditions:
  Condition 1: Standing with standardized flat shoes. Perform three trials for each participant. Calculate and record the mean as baseline data. Condition 2: Standing with a standardized heel lift insole inside the flat shoes.
  Conduct three trials. Record the mean for comparative analysis.
Diagnostic Test: Photograph participants from anterior and lateral views to assess knee valgus angle and lumbosacral angle. — Capture two sets of photographs for each participant:
  Set 1: Wearing flat shoes. Set 2: Wearing the heel lift insole inside the flat shoes. Compare knee valgus angle and lumbosacral angle under both conditions. Ensure consistency and reliability by following standardized protocols and performing repeated measurements.
  Analyze the effects of heel lift insoles on muscle activity and postural alignment.

SUMMARY:
This observational study aims to investigate the effect of heel lift insole on kinematics and kinetics of the lower limb and lumbar spine among healthy individuals.

DETAILED DESCRIPTION:
This clinical trial will be conducted among physiotherapy students at Misr University for Science and Technology. Participants will be recruited based on predefined inclusion criteria, and informed consent will be obtained prior to their involvement. Once enrolled, each participant will complete a standardized demographic questionnaire and undergo height and weight measurements to calculate their Body Mass Index (BMI). Those with BMI values outside the normal range, as defined by Shrestha et al. (2023), will be excluded to reduce confounding factors.

Before testing begins, participants will be familiarized with all equipment and procedures. Electromyographic (EMG) data will then be collected to measure maximum muscle activity in the bilateral erector spinae, rectus femoris, and both medial and lateral gastrocnemius muscles. EMG measurements will be taken under two conditions: first, while standing in standardized flat shoes, and second, while wearing a standardized heel lift insole inside the same shoes. Three trials will be performed in each condition, and the mean amplitude will be used for analysis.

In addition to EMG, kinematic data will be assessed using Kinovea software. Photographs will be captured from anterior and lateral views to evaluate each participant's Q angle and lumbosacral angle. As with EMG, these measurements will be repeated under both footwear conditions (flat shoes alone and flat shoes with heel lift insoles), and the results will be compared.

All procedures will follow standardized protocols to ensure consistency and reliability. The primary outcome measure is muscle activity (maximum EMG amplitude), while secondary outcomes include changes in the Q-angle and lumbosacral angle. The study aims to evaluate the impact of heel lift insoles on lower limb muscle activity and postural alignment in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult non-athletic individuals with age range between (18: 25) years old (Joshi et al., 2024).
* Height between (160 - 180 cm).
* Body mass index between (18.5:24.99) Kg/ m² (Joshi et al., 2024).
* Foot length between (23,3 - 28.0 cm).
* Never used heel lift insole.
* Participants must have a normal and pain-free range of motion in the lower limbs and spine (Hapsari et al., 2016).
* Participants must demonstrate stable balance and coordination in weight-bearing activities (Hapsari et al., 2016).

Exclusion Criteria:

* Traumatic conditions of the lower limb (Joshi et al., 2024).
* Pelvis and lower limb musculoskeletal disorders (Joshi et al., 2024).
* Previous orthopedic disorders or neurological deficit of the lower limb (Joshi et al., 2024).
* Previous surgery of the lower limbs (Lindenberg et al., 2019).
* Any sensory problems.
* Neuromuscular diseases such as multiple sclerosis, intervertebral disc disorders…etc (Joshi et al., 2024).
* Pregnancy.
* Cancer Patients.
* Immunodeficiency diseases.
* Psychological disorders (depression - anxiety).
* Chronic diseases as (diabetes - hypertension).
* Participants with lower limbs deformity (Joshi et al., 2024).
* Participants with specific lower limb muscles weakness.
* Low back pain in the past 30 days (Colonna et al., 2024).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Individuals
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Muscle activity (Maximum amplitude in microvolt) - Electromyography Device Using interference pattern | 3 Months

SECONDARY OUTCOMES:
Q-Angle using objective Kinovea 2D software | 3 months
Lumbo-Sacral Angle using objective Kinovea 2D software | 3 Months

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Misr University for science and technology, Giza, Giza Governorate
  - Misr University for science and technology, Physical Therapy College, EMG and NCV Lab, Giza

IPD SHARING:
Plan to Share IPD: No